CLINICAL TRIAL: NCT00348764
Title: Treatment of Greater Saphenous Vein (GSV) Insufficiency Using Echo-Guided Sclerotherapy With Lauromacrogol 400 Foam -Comparative Study of 3% Versus 1% Concentration.
Brief Title: ESGVS: Sclerotherapy With Lauromacrogol
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University Hospital, Grenoble (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: DCIC 03 38
Record Dates: First submitted 2006-07-05; First posted 2006-07-06 (Estimated); Last update posted 2006-07-06 (Estimated); Status verified 2006-07

CONDITIONS: Venous Insufficiency; Saphenous Vein
Keywords: lauromacrogol; Sclerotherapy
MeSH Terms: conditions — Venous Insufficiency | interventions — Polidocanol

INTERVENTIONS:
Drug: lauromacrogol

SUMMARY:
To evaluate the efficacy and the tolerance of echoguided sclerotherapy using Lauromacrogol 400 foam for the treatment of Great Saphenous Vein (GSV) insufficiency. A comparative study of 3% versus 1% Lauromacrogol 400 foam.

DETAILED DESCRIPTION:
A multicenter randomized double blind study to evaluate the efficacy and the tolerance of echoguided sclerotherapy using 3% versus 1% Lauromacrogol 400 foam in the treatment of Great Saphenous Vein (GSV) insufficiency.

One hundred fifty eligible patients will be recruited during 6 months from 9 study centers with a follow up period of 3 years and 7 visits at day 8, 6 weeks, 3 months, 6 months, 1,2 ,and 3 years.

After randomization, the patients will be treated by echoguided sclerotherapy with 1% or 3% Lauromacrogol 400 foam (ratio 1:1).

Monitoring is performed by doppler at 8 days, 6 weeks, 6 months , 1,2 ,and 3 years.

Effectiveness of sclerotherapy is determined at 6 weeks, 3 months and 6 months. A additional injection of 4 ml of foam can be performed if needed.

Severity clinical score and Quality-of-life questionnaire are performed at 6 months ,1 ,2, and 3 years.

The absence of obliteration with a reflux of crural great saphenous vein at 6 months will be a criterion of therapeutic failure.

The therapeutic success or failure criteria are evaluated by a non investigator angiologist for 5 patients randomized from each investigational site at 1, 2 and 3 years.

ELIGIBILITY:
Inclusion Criteria:

* 25 - 75 years
* Hawaii CEAP classification : C2-5 Ep, As2-3 Pr
* Clinical Varicose veins C2, Edema C3, Skin changes C4, Healed ulcer C5
* Etiology Ep Primary GSV insufficiency
* As2-3: Ostial and or crural truncular GVS incompetence
* Maximal inferior diameter of the leg GSV (patient in decubitus) between 4 and 8mm
* Pr: reflux by echo doppler in orthostatism > 1 second
* Information consent form signed by the investigator and the patient.

Exclusion Criteria:

* deep venous reflux (CEAP: Ad)
* Short saphenous vein or non saphenous network insufficiency (CEAP: A4-5)
* Clinical class: C1 or C6
* Recurrent GSV varicose veins after stripping
* Thrombophilia or antecedent of deep vein thrombosis
* Psychiatric disorders
* Known allergy to Lauromacrogol or to one of its component
* Arteriopathy. (IPS < 0.8)
* Post-thrombotic disease
* Chronic hepatoma
* Renal insufficiency (creatinine > 150 micromol/l)

Ages: 25 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150
Dates: Start 2004-03; Study Completion 2006-12

PRIMARY OUTCOMES:
Removal of truncular GSV incompetence evaluated at 6 months by echo doppler: no persistence of "sus gonal" saphenous reflux > 1 second.

SECONDARY OUTCOMES:
Removal of truncular GSV incompetence evaluated at 6 months by echo doppler: no persistence of "sus gonal" saphenous reflux > 1 second.

CONTACTS AND LOCATIONS:
Overall Officials: DIAMAND Jean Marc, Principal Investigator — Institut National de la Santé Et de la Recherche Médicale, France
Locations (1):
- Center of Vascular Medecine - 7 rue Lesdiguières, Grenoble, France

REFERENCES:
- [Background] Bosson JL, Riachi M, Pichot O, Michoud E, Carpentier PH, Franco A. Diameters of acute proximal and distal deep venous thrombosis of the lower limbs. Int Angiol. 1998 Dec;17(4):260-7. PMID 10204659
- [Background] Ferretti GR, Bosson JL, Buffaz PD, Ayanian D, Pison C, Blanc F, Carpentier F, Carpentier P, Coulomb M. Acute pulmonary embolism: role of helical CT in 164 patients with intermediate probability at ventilation-perfusion scintigraphy and normal results at duplex US of the legs. Radiology. 1997 Nov;205(2):453-8. doi: 10.1148/radiology.205.2.9356628.
- [Background] Barro C, Bosson JL, Pernod G, Carpentier PH, Polack B. Plasma D-dimer testing improves the management of thromboembolic disease in hospitalized patients. Thromb Res. 1999 Sep 1;95(5):263-9. doi: 10.1016/s0049-3848(99)00042-0. No abstract available. PMID 10515291
- [Background] Bosson JL, Labarere J, Sevestre MA, Belmin J, Beyssier L, Elias A, Franco A, Le Roux P. Deep vein thrombosis in elderly patients hospitalized in subacute care facilities: a multicenter cross-sectional study of risk factors, prophylaxis, and prevalence. Arch Intern Med. 2003 Nov 24;163(21):2613-8. doi: 10.1001/archinte.163.21.2613. PMID 14638561
- [Background] Bosson JL, Labarere J, Barrellier MT, Belmin J, Couturier P, Le Roux P, Sevestre MA; Association pour la Promotion de l'Angiologie Hospitaliere (APAH). [Practice guidelines for the prevention of venous thromboembolism in elderly patients hospitalized in subacute care and rehabilitation facilities (short text). Association for the Promotion of Hospital Angiology]. J Mal Vasc. 2003 Oct;28(4):209-18. No abstract available. French. PMID 14618112